CLINICAL TRIAL: NCT03722472
Title: A Phase 1, Double-Blind, Randomized Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of the Single-Vial Lyophilized ID93 + GLA-SE Vaccine Administered Intramuscularly in Healthy Adult Subjects
Brief Title: Phase 1 Clinical Trial of Single-Vial ID93 + GLA-SE in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IDRI-TBVPX-120; DMID 17-0104 (Other: NIH/NIAID/DMID); 272201400041C-0-0-1 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary TB
Keywords: Vaccine, recombinant, adjuvant, GLA-SE, ID93
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All clinical staff and the participants are blinded to treatment, with the exception of the clinical pharmacist who prepares the vaccines and syringes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single-vial ID93 + GLA-SE (Experimental): Single-vial presentation of ID93 + GLA-SE. Participants will receive two intramuscular (IM) injections of the vaccine on Days 0 and 56. 2 mcg ID93 and 5 mcg GLA-SE in 0.5 mL volume will be given per injection.
  Interventions: Biological: ID93 + GLA-SE
- Two-vial ID93 + GLA-SE (Active Comparator): Two-vial presentation of ID93 + GLA-SE. Participants will receive two intramuscular (IM) injections of the vaccine on Days 0 and 56. 2 mcg ID93 and 5 mcg GLA-SE in 0.5 mL volume will be given per injection.
  Interventions: Biological: ID93 + GLA-SE

INTERVENTIONS:
Biological: ID93 + GLA-SE — The single-vial lyophilized vaccine will be reconstituted with WFI. For the two-vial presentation, the lyophilized ID93 will be reconstituted with WFI and mixed with liquid GLA-SE.

SUMMARY:
This is a phase 1, double-blind, randomized clinical trial to evaluate the safety, tolerability, and immunogenicity of single-vial lyophilized ID93 + GLA-SE compared to the two-vial presentation consisting of lyophilized ID93 and liquid GLA-SE administered as two IM injections in healthy adult subjects (aged 18 - 55).

DETAILED DESCRIPTION:
Subjects will receive a total of two doses administered IM on Days 0 and 56. Subjects will be monitored for approximately 421 days (one year following the last study injection), including safety laboratory analyses done just prior to and 7 days following each study injection. Tears and nasal swabs will be obtained for exploratory antibody analysis at Days 0, 70, and 224. Blood samples will be obtained for immunological assays (secondary and exploratory) at Days 0, 7, 14, 56, 63, 70, 84, and 224).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 to 55 years of age.
2. In good general health as confirmed by a medical history and physical exam, vital signs*, and screening laboratories conducted no more than 30 days prior to study injection administration.

   *Temperature <38°C, respiratory rate < 17 breaths pm, heart rate ≤100 bpm and >54 bpm, systolic blood pressure ≤140 mmHg and >89 mmHg, diastolic blood pressure ≤90 mmHg and ≥60 mmHg.

   NOTE: Athletically trained subjects with a pulse ≥40 may be enrolled at the discretion of the principal investigator or designated licensed clinical investigator.
3. Screening laboratory values within normal limits: sodium, potassium, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, random glucose, total WBC count, hemoglobin, and platelet count.
4. Negative HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
5. Urine dipstick for protein and glucose (negative to trace protein are acceptable).
6. Women of childbearing potential* in sexual relationships with men must agree to practice acceptable contraception** for the 30-day period before Day 0 through 90 days after the last study injection.

   *Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal). Post-menopausal defined as at least 12 months spontaneous amenorrhea and confirmed with FSH > 40 mIU/ml.

   **Includes, but is not limited to, sexual abstinence, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject receiving study product, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing ®, and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
7. Able to understand and comply with planned study procedures and willing to be available for all study-required procedures, visits and calls for the duration of the study.
8. Provide written informed consent before initiation of any study procedures.
9. Willing to abstain from donating whole blood or blood derivatives until 90 days after the final study injection.

Exclusion Criteria:

1. Previous exposure to ID93 vaccines or experimental products containing GLA-SE.
2. History of treatment for active or latent tuberculosis infection.
3. History or evidence of active or documented latent tuberculosis, or positive QuantiFERON®-TB Gold test.
4. Shared a residence within the last year prior to randomization with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis.
5. Received a tuberculin skin test within 3 months (90 days) prior to randomization.
6. History of autoimmune disease or immunosuppression.
7. Used immunosuppressive medication (e.g., oral or injected steroids) within 3 months prior to randomization (inhaled and topical corticosteroids are permitted).
8. Received any investigational drug therapy or investigational vaccine within past 6 months prior to randomization, or planned participation in any other investigational study during the study period.
9. Received investigational TB vaccine at any time prior to randomization.
10. Received any vaccine within 30 days prior to the first study vaccination and no planned immunizations between Day 0-84 or Day 210-224 due to the washout period prior to immunology blood draws.
11. History or laboratory evidence of immunodeficiency state including but not limited to laboratory indication of HIV-1 infection at screening.
12. History of allergic disease or reactions, likely to be exacerbated by any component of the study vaccine.
13. History of allergic reaction to kanamycin-related antibiotics.
14. Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines or unknown allergens.
15. Previous medical history that may compromise the safety of the subject in the study, including but not limited to: severe impairment of pulmonary function from tuberculosis infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; or uncontrolled epilepsy or infantile spasms.
16. Known or suspected alcohol or drug abuse within the past 5 years.
17. Smokes 1 pack or more of cigarettes per day.
18. History of keloid formation or excessive scarring.
19. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine, including axillary lymphadenopathy.
20. Received a blood transfusion or immunoglobulin within the past 3 months prior to randomization.
21. Donated blood products (platelets, whole blood, plasma, etc.) within past 1 month prior to randomization.
22. Presence of any febrile illness, oral temperature of >100.4 °F/38.0 °C within 24 hours of study injection administration. Such subjects may be re-evaluated for enrolment after resolution of illness.
23. Positive serum (at screening visit only) or urine pregnancy test at screening or within 24 hours prior to study injection for women of childbearing potential.
24. Breastfeeding at any time throughout the study.
25. Rash, tattoos, or any other dermatological condition on the upper anterolateral arm that could adversely affect the vaccine injection site or interfere with its evaluation.
26. BMI <18 or >35 kg/m2.
27. Any medical or neuropsychiatric condition which, in the Investigator's opinion, would render the subject incompetent to provide informed consent or unable to provide valid safety observations and reporting.
28. Cancer or treatment for cancer within 3 years of study injection administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible.
29. Subjects unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Fox, PhD, Principal Investigator — Access to Advanced Health Institute (AAHI)
Locations (1):
- Saint Louis University - Center for Vaccine Development, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sagawa ZK, Goman C, Frevol A, Blazevic A, Tennant J, Fisher B, Day T, Jackson S, Lemiale F, Toussaint L, Kalisz I, Jiang J, Ondrejcek L, Mohamath R, Vergara J, Lew A, Beckmann AM, Casper C, Hoft DF, Fox CB. Safety and immunogenicity of a thermostable ID93 + GLA-SE tuberculosis vaccine candidate in healthy adults. Nat Commun. 2023 Mar 6;14(1):1138. doi: 10.1038/s41467-023-36789-2. PMID 36878897
- See also: Safety and immunogenicity of a thermostable ID93 + GLA-SE tuberculosis vaccine candidate in healthy adults — http://www.nature.com/articles/s41467-023-36789-2

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-vial Presentation ID93 + GLA-SE: Thermostable lyophilized single-vial presentation of ID93 + GLA-SE (2 µg ID93, 5 µg GLA) given as two intramuscular (IM) injections on Days 0 and 56.
- Two-vial Presentation ID93 + GLA-SE: Non-thermostable two-vial presentation of ID93 (2 µg, lyophilized) + GLA-SE (5 µg, liquid) given as two intramuscular (IM) injections on Days 0 and 56.
Period: Overall Study
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Started | 23 | 25
Completed | 23 | 22
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: males and females, ages 18-55 inclusive
Groups:
- Single-vial Presentation ID93 + GLA-SE: ID93 + GLA-SE (2 µg ID93, 5 µg GLA) [lyophilized, single-vial] given as two intramuscular (IM) injections on Days 0 and 56.
- Two-vial Presentation ID93 + GLA-SE: ID93 (2 µg, lyophilized) + GLA-SE (5 µg, liquid) [two-vial presentation] given as two intramuscular (IM) injections on Days 0 and 56.
- Total: Total of all reporting groups
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 23 | 43
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Local Injection Site Reactogenicity
Description: The number of subjects experiencing solicited local injection site reactions within 7 days following each study injection.
Time Frame: 7 days following each injection
Population: Safety population (n=48). All subjects receiving at least one study injection.
Measure: Number; unit: participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
participants | 22 | 21

2. Primary Outcome: Systemic Reactogenicity
Description: The number of subjects experiencing solicited systemic reactions within 7 days following each study injection.
Time Frame: 7 days following each injection
Population: Safety population (n=48). All subjects receiving at least one study injection.
Measure: Number; unit: participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
participants | 9 | 12

3. Primary Outcome: All Adverse Events
Description: The number of subjects spontaneously reporting adverse events from Day 0 through Day 84.
Time Frame: Day 0 - 84
Population: Safety population (n=48). All subjects received at least one study injection.
Measure: Number; unit: participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
participants | 23 | 24

4. Primary Outcome: Serious Adverse Events
Description: The number of serious adverse events considered related to any of the study injections reported at any point during the study period.
Time Frame: Day 0 - 421
Population: Safety population (n=48). All subjects received at least one study injection.
Measure: Number; unit: participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
participants | 0 | 0

5. Secondary Outcome: IgG Antibody Response Rate
Description: Total IgG antibody ELISA: Responder rate is defined as the proportion of subjects with at least a 4-fold increase from baseline in IgG antibody titer for ID93 antigen.
Time Frame: Days 0, 14, 56, 70, 84, and 224
Population: Immunogenicity population: all eligible subjects who have received at least one study injection, for whom data concerning post-baseline immunogenicity endpoint measures are available, and major protocol deviations are absent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
percentage of participants
  Day 14 Responder rate: number analyzed (Participants) | 23 | 24
  Day 14 Responder rate | 30.4 [13.21 to 52.92] | 25.0 [9.77 to 46.71]
  Day 56 Responder rate: number analyzed (Participants) | 23 | 22
  Day 56 Responder rate | 60.9 [38.54 to 80.29] | 40.9 [20.71 to 63.65]
  Day 70 Responder rate: number analyzed (Participants) | 23 | 22
  Day 70 Responder rate | 100 [85.18 to 100.0] | 90.9 [70.84 to 98.88]
  Day 84 Responder rate: number analyzed (Participants) | 22 | 22
  Day 84 Responder rate | 90.9 [70.84 to 98.88] | 95.5 [77.16 to 99.88]
  Day 224 Responder rate: number analyzed (Participants) | 20 | 22
  Day 224 Responder rate | 85.0 [62.11 to 96.79] | 63.6 [40.66 to 82.80]

6. Secondary Outcome: IgG Antibody Response Magnitude
Description: Total IgG mean endpoint titer for ID93
Time Frame: Days 0, 14, 56, 70, 84, and 224
Population: All subjects who have received at least one study injection, for whom data concerning post-baseline immunogenicity endpoint measures are available, and major protocol deviations are absent.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
titer
  Day 0 Geometric Mean MEPT | 57 [49 to 66] | 74 [45 to 123]
  Day 14 Geometric Mean MEPT: number analyzed (Participants) | 23 | 24
  Day 14 Geometric Mean MEPT | 147 [83 to 260] | 140 [94 to 209]
  Day 56 Geometric Mean MEPT: number analyzed (Participants) | 23 | 22
  Day 56 Geometric Mean MEPT | 250 [154 to 405] | 259 [126 to 530]
  Day 70 Geometric Mean MEPT: number analyzed (Participants) | 23 | 22
  Day 70 Geometric Mean MEPT | 10868 [5971 to 19780] | 2583 [1608 to 4147]
  Day 84 Geometric Mean MEPT: number analyzed (Participants) | 22 | 22
  Day 84 Geometric Mean MEPT | 5592 [2753 to 11362] | 2522 [1711 to 3716]
  Day 224 Geometric Mean MEPT: number analyzed (Participants) | 20 | 22
  Day 224 Geometric Mean MEPT | 913 [510 to 1634] | 445 [273 to 726]

7. Secondary Outcome: Cytokine Response
Description: PBMC ELISpot: IFN-γ response to the ID93 antigen. Responder status is determined by the SCHARP method.
Time Frame: Days 0, 14, 56, 70, 84, and 224
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
percentage of participants
  Day 0 Responder rate | 13.0 [2.78 to 33.59] | 20.0 [6.83 to 40.70]
  Day 14 Responder rate: number analyzed (Participants) | 22 | 25
  Day 14 Responder rate | 45.5 [24.39 to 67.79] | 32.0 [14.95 to 53.5]
  Day 56 Responder rate: number analyzed (Participants) | 23 | 22
  Day 56 Responder rate | 34.8 [16.38 to 57.27] | 31.8 [13.86 to 54.87]
  Day 70 Responder rate: number analyzed (Participants) | 23 | 21
  Day 70 Responder rate | 69.6 [47.08 to 86.79] | 76.2 [52.83 to 91.79]
  DAY 84 Responder rate: number analyzed (Participants) | 22 | 21
  DAY 84 Responder rate | 68.2 [45.13 to 86.14] | 66.7 [43.03 to 85.41]
  Day 224 Responder rate: number analyzed (Participants) | 20 | 19
  Day 224 Responder rate | 65 [40.78 to 84.61] | 52.6 [28.86 to 75.55]

8. Secondary Outcome: Cytokine Response
Description: PBMC ELISpot: IL-10 response to the ID93 antigen. Responder status is determined by the SCHARP method.
Time Frame: Days 0, 14, 56, 70, 84 and 224
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
percentage of participants
  Day 0 Responder rate | 4.3 [0.11 to 21.95] | 8.0 [0.98 to 26.03]
  Day 14 Responder rate: number analyzed (Participants) | 22 | 23
  Day 14 Responder rate | 0 [0.00 to 15.44] | 4.3 [0.11 to 21.95]
  Day 56 Responder rate: number analyzed (Participants) | 23 | 22
  Day 56 Responder rate | 4.3 [0.11 to 21.95] | 4.5 [0.12 to 22.84]
  Day 70 Responder rate: number analyzed (Participants) | 23 | 20
  Day 70 Responder rate | 30.4 [13.21 to 52.92] | 0 [0.00 to 16.84]
  Day 84 Responder rate: number analyzed (Participants) | 22 | 19
  Day 84 Responder rate | 18.2 [5.19 to 40.28] | 10.5 [1.30 to 33.14]
  Day 224 Responder rate: number analyzed (Participants) | 20 | 18
  Day 224 Responder rate | 10.0 [1.23 to 31.70] | 0 [0.00 to 18.53]

9. Secondary Outcome: T Cell Response
Description: PBMC ICS: Responder Rate of the "Any Two" CD4 T cell responses to the ID93 antigen; CD4 T cells producing 1 or more cytokines (IFN-γ, TNF, IL-2, IL-4, IL-21 and CD154) simultaneously in response to stimulation with the ID93 antigen as measured by intracellular cytokine staining of PBMCs.
Time Frame: Days 0, 7, 14, 56, 63, 70, 84 and 224
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
percentage of participants
  Day 0 Responder rate | 4.3 [0.11 to 21.95] | 4.0 [0.10 to 20.35]
  Day 7 Responder rate: number analyzed (Participants) | 21 | 25
  Day 7 Responder rate | 4.8 [0.12 to 23.82] | 4.0 [0.10 to 20.35]
  Day 14 Responder rate: number analyzed (Participants) | 20 | 24
  Day 14 Responder rate | 15.0 [3.21 to 37.89] | 4.2 [0.11 to 21.12]
  Day 56 Responder rate: number analyzed (Participants) | 22 | 20
  Day 56 Responder rate | 13.6 [2.91 to 34.91] | 0 [0.00 to 16.84]
  Day 63 Responder rate: number analyzed (Participants) | 22 | 22
  Day 63 Responder rate | 36.4 [17.20 to 59.34] | 13.6 [2.91 to 34.91]
  Day 70 Responder rate: number analyzed (Participants) | 22 | 21
  Day 70 Responder rate | 59.1 [36.35 to 79.29] | 38.1 [18.11 to 61.56]
  Day 84 Responder rate: number analyzed (Participants) | 20 | 20
  Day 84 Responder rate | 50.0 [27.20 to 72.80] | 30.0 [11.89 to 54.28]
  Day 224 Responder rate: number analyzed (Participants) | 16 | 19
  Day 224 Responder rate | 31.3 [11.02 to 58.66] | 26.3 [9.15 to 51.20]

10. Secondary Outcome: T Cell Response
Description: PBMC ICS: Responder Rate of the "Any Two" CD8 T cell responses to the ID93 antigen; CD8 T cells producing 1 or more cytokines (IFN-γ, TNF, IL-2, IL-4, IL-21 and CD154) simultaneously in response to stimulation with the ID93 antigen as measured by intracellular cytokine staining of PBMCs.
Time Frame: Days 0, 7, 14, 56, 63, 70, 84 and 224.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
Number analyzed (Participants) | 23 | 25
percentage of participants
  Day 0 Responder rate | 0 [0.00 to 14.82] | 0 [0.00 to 13.72]
  Day 7 Responder rate: number analyzed (Participants) | 21 | 25
  Day 7 Responder rate | 4.8 [0.12 to 23.82] | 0 [0.00 to 13.72]
  Day 14 Responder rate: number analyzed (Participants) | 20 | 24
  Day 14 Responder rate | 15.0 [3.21 to 37.89] | 0 [0.00 to 14.25]
  Day 56 Responder rate: number analyzed (Participants) | 22 | 20
  Day 56 Responder rate | 4.5 [0.12 to 22.84] | 0 [0.00 to 16.84]
  Day 63 Responder rate: number analyzed (Participants) | 22 | 22
  Day 63 Responder rate | 4.5 [0.12 to 22.84] | 9.1 [1.12 to 29.16]
  Day 70 Responder rate: number analyzed (Participants) | 22 | 21
  Day 70 Responder rate | 0 [0.00 to 15.44] | 4.8 [0.12 to 23.82]
  Day 84 Responder rate: number analyzed (Participants) | 20 | 20
  Day 84 Responder rate | 0 [0.00 to 16.84] | 5.0 [0.13 to 24.87]
  Day 224 Responder rate: number analyzed (Participants) | 16 | 19
  Day 224 Responder rate | 6.3 [0.16 to 30.23] | 15.8 [3.38 to 39.58]

ADVERSE EVENTS:
Time Frame: 421 days
Description: Solicited adverse events within 7 days and unsolicited adverse events within 28 days after each study injection; serious adverse events (SAEs) and potential immune-mediated medical conditions (PIMMCs) after the first study injection until end of study follow-up.
Arm/Group | Single-vial Presentation ID93 + GLA-SE | Two-vial Presentation ID93 + GLA-SE
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 23/23 | 24/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-vial Presentation ID93 + GLA-SE (N=23) | Two-vial Presentation ID93 + GLA-SE (N=25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 — Injection related reactions
Fatigue (General disorders) | 6 | 10 — Injection related reactions
Headache (Nervous system disorders) | 4 | 7 — Injection related reactions
Injection site pain (General disorders) | 22 | 21 — Injection related reactions
Injection site induration (General disorders) | 3 | 0 — Injection related reactions
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5 — Injection related reactions
Haemoglobin decreased (Investigations) | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT03722472/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT03722472/SAP_001.pdf